CLINICAL TRIAL: NCT06910527
Title: Study of the Evolution of Circulating Plasma and Urinary DNA of Renal Origin in Kidney Transplant Patients
Brief Title: Study of the Plasma and Urinary cfDNA of in Kidney Transplant Patients
Acronym: PLAKID-TRANSP
Status: Recruiting | Type: Observational
Sponsor: Poulet Geoffroy (Industry)
Collaborators: University Hospital, Rouen (Other)
Responsible Party: Sponsor-Investigator, Poulet Geoffroy, Doctor, CGenetix
Organization: CGenetix (Industry)
Other Study IDs: PLAKID-TRANSP
Record Dates: First submitted 2025-03-19; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Transplant Rejection; Transplant Kidney
Keywords: Kidney transplantation; Cell-free DNA; Epigenetic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and urine sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Kidney transplant patient eligible to a kidney biopsy: Kidney transplant patient eligible to a kidney biopsy (protocol and indication biopsy)

SUMMARY:
It has been shown that the amount of circulating donor-cell-free DNA increases in patients with transplant rejection. Quantification of single nucleotide polymorphisms (SNPs) present in circulating donor DNA currently allows for early identification of transplant rejection, but not for characterization, i.e., identification of the affected renal fraction of the graft.

Recently, in healthy subjects, teams have shown that it is possible to identify the tissue origin of donor-cell-free DNA, based on the epigenetic properties of circulating DNA.

CGenetix is a MedTech company developing an in vitro diagnostic medical device to identify and quantify kidney graft degradation during transplant rejection. The objective of this study is to evaluate the sensitivity of the proposed technology to detect circulating renal DNA released into the blood and urine in kidney transplant patients with or without graft rejection.

DETAILED DESCRIPTION:
Screening Step :

As part of routine kidney transplant patient monitoring, humoral or cellular rejection may be suspected when graft function deteriorates, proteinuria increases, or antibodies against the graft appear. If rejection is suspected, and in the absence of contraindications, a graft biopsy is scheduled during a conventional inpatient or midweek hospitalization to perform a pathological examination.

Inclusion Step :

1. Transplant patient follow-up stage - Nephrology-transplant consultation: Scheduling of a graft biopsy for suspected rejection.
2. Patient inclusion stage in the study, corresponding to the day the solid biopsy is performed in a conventional or day hospitalization setting.
3. The patient's signature of the non-objection notice and blood samples for the research to be conducted can be taken on the same day. A minimum reflection period of 6 hours has been decided for this study to allow the patient to participate in the study.

During the patient inclusion stage, a non-objection notice and written, free consent for participation in the study and the collection of biological samples signed by the patient will be collected by the coordinating investigator or the physician (declared to be trained in research). A minimum reflection period of 6 hours was set before proposing to the patient to participate in the study.

Admission of patients to the Nephrology-Transplantation Department for suspected rejection

Within 24 hours prior to the biopsy for:

* Two PAXgene Blood ccfDNA Tubes (100) - (Cat. No. / ID: 768115; Beckson Dickinson) containing 10 mL of blood in addition to the blood sample taken as part of the treatment will be collected.
* One 20 mL urine container (Urine Collection Bottle, Non-Sterile, 500 pieces; Item No.: 128139; Praxisdienst) supplemented with a preservative agent "Streck® Urine Preserve 12 x 5.0 mL; Item No. 230599: Eurobio Scientific") in addition to the urine sample taken as part of the treatment will be collected.

These two additional blood tubes and one urine container for research purposes will be collected weekly by an authorized carrier for analysis at CGenetix. Raw urine and blood samples will be stored at room temperature in the Nephrology-Transplantation Department of Rouen University Hospital.

The urine tubes and containers will be centrifuged, and the plasma and urine supernatants will be frozen in cryovials at -80°C at CGenetix for analysis.

Biological Collection Plasma and urine samples collected for the specific purposes of the research will not be included in a biological collection. They will be used entirely for the purposes of this research.

During the research, the samples in the collection will be stored at the CGenetix laboratory located at 4 rue Pierre Fontaine, EVRY-COURCOURONNES, 91058, under the responsibility of its president, Geoffroy POULET.

Study duration : 24 months Rouen University Hospital performs an average of 140 renal biopsies annually. Among these patients, it is estimated that 10% of these biopsies are humoral rejections and 10% are cellular rejections.

Data collection Modality Data collection will be conducted by the principal investigator, Dr. Tristan DE NATTES, via the Rouen University Hospital's electronic medical records, using CDP2 software for the histological and biological data components within the Rouen University Hospital's Nephrology-Transplantation Department.

Biological results will be obtained from blood and urine samples collected as part of routine care upon the patient's inclusion in the study: blood electrolytes, creatinine, proteinuria, hematuria, and leukocyturia just before the renal biopsy (RBB) is performed.

The histological data (score determined according to the Banff classification and pathology report) will be those collected from the reading of the renal biopsy by the Rouen University Hospital's pathologists.

No clinical data will be collected from the patient's medical records in this study. The data collected in this study (listed in Addendum No. 2: List of Data Collected in This Study) will be pseudo-anonymized by the Rouen University Hospital and will only be transferred from the Rouen University Hospital to the company CGenetix. The data will not be transferred outside of France. The Rouen University Hospital is responsible for the pseudo-anonymization of patient data received in their hospital department.

This data will be collected in a password-protected Excel database hosted on a computer in the Rouen University Hospital Kidney Transplantation Department, which is itself password-protected and to which only Dr. Tristan DE NATTES and the clinical research associates of the Nephrology Department will have access. A correspondence table will be created by the principal investigator between patient identities and their research identification numbers. This file will be stored in a password-protected Excel file hosted on a computer in the Kidney Transplantation Department of Rouen University Hospital, which is password-protected and accessible only by Dr. Tristan de NATTES.

The circulating renal biomarker data tested in this research protocol will be generated by CGenetix and collected in a password-protected Excel file hosted on a computer in CGenetix's R&D department, which is password-protected and accessible only by the study's scientific director, Dr. Geoffroy Poulet, and CGenetix's statistician, Mr. Thomas Bersez. After transmission of the biological and histological data collection table from Rouen University Hospital to CGenetix, the circulating renal biomarker data will be compiled into a single Excel file and placed on a secure, HDS-certified Dropbox server within CGenetix, to which only the principal investigator, Dr. Tristan DE NATTES, the study's scientific director, Dr. Geoffroy POULET, and CGenetix's statistical director, Mr. Thomas BERSEZ, will have access.

The principal investigator and the clinical research associates assigned to this study will take all necessary precautions to ensure the confidentiality of information relating to the research, the individuals participating in it, particularly with regard to their identity, and the results obtained. These individuals, like the investigators themselves, are subject to professional secrecy (in accordance with the conditions defined by Articles 226-13 and 226-14 of the French Criminal Code). During and after the research involving human subjects, the data collected on the subjects and transmitted to the sponsor by the investigators (or any other specialized personnel) will be made non-identifying. Under no circumstances should the data clearly display the names of the subjects concerned or their addresses. Only the initials of the first and last names will be recorded, along with a coded number specific to the research indicating the order of inclusion of the subjects.

The sponsor will ensure that each person participating in the research has given their consent for access to the individual data concerning them, which is strictly necessary for the quality control of the research.

Data flow The data will be collected by the research team and the principal investigator in a pseudo-anonymized form in a password-protected Excel file hosted on the hospital network.

The biological and histological data collection table listed in section 6.1 is then transferred to CGenetix via a secure Dropbox link, accessible only by the principal investigator at Rouen University Hospital, the CGenetix scientific director, and the CGenetix statistician. This transmission of the biological and histological data collection table will be carried out in batches for every 30 patients included in the study. CGenetix hosts this data both on the study's scientific director's computer and on a secure, HDS-certified Dropbox server. The sponsor CGenetix, using the correspondence table and the patient biological and histological data collection table, will compile the quantification data for circulating renal biomarkers into the collection table to create a consistent file and consistent data for statistical analysis.

• Renal degradation biomarker data generated by CGenetix The renal degradation biomarker data (total kidney, tubular, and vascular) are generated within CGenetix using its analytical pipeline. The data is stored in a secure database on the study's scientific director's computer and also on a secure cloud dedicated to the management of sensitive data, certified ISO 27001, 27017, 27018, 27701, and HDS. The clinical data from the care collected by the Rouen University Hospital and included in the statistical analysis of the clinical study are also stored on the computer of the scientific manager of the study and on the cloud (secure Dropbox space) of the company CGenetix.

ELIGIBILITY:
Inclusion Criteria:

* Patients living with a kidney transplant
* Admitted for suspected transplant rejection requiring a renal biopsy (RBB) as an indication

Exclusion Criteria:

* Patients with cognitive and mental disorders rendering them unable to express their non-opposition to participation in the study
* Not covered by a social security system.
* Under guardianship or guardianship, or under legal protection.
* Patients who have expressed their refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients living with a kidney transplant eligible for a protocol biopsy or indication for suspected graft rejection
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-05-30 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Renal cell-free DNA in plasma and urine | 24 Hours
  Quantification of Renal-cell-free DNA in plasma and urine exprimed in copy / mL of biological fluid

CONTACTS AND LOCATIONS:
Overall Officials: Geoffroy GP POULET, PhD, Study Director — CGenetix; TRISTAN DE NATTES, MEDICAL DOCTOR, Principal Investigator — CHU ROUEN UNIVERSITY
Locations (1):
- Chu Rouen-Bois Guillaume, Rouen, France

IPD SHARING:
Plan to Share IPD: No